CLINICAL TRIAL: NCT06122844
Title: Feasibility of Mindfulness-based Training for Teachers and Young Children for Social Emotional and Ethical Development (SEED)
Brief Title: Social Emotional and Ethical Development (SEED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Xi'an Jiaotong-Liverpool University (Unknown)
Responsible Party: Principal Investigator, Winnie W.S. MAK, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SBRE-22-0785A
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-05

CONDITIONS: Development, Child; Mindfulness; Mental Well-being
Keywords: Social, Emotional, and Ethical Development; Mindfulness; Mental well-being; Young children
MeSH Terms: conditions — Psychological Well-Being | interventions — Seeds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Social, Emotional, and Ethical Development (SEED) curriculum (Experimental): The kindergartens, teachers, and children will receive the training and SEED curriculum. Upon informed consent from the school principals and parents, parents, teachers, and children will complete pre-, post-, and 4-week follow-up assessments. Focus group interviews will be conducted with teachers to understand their acceptability, demand, practicality, integration, and efficacy of the teacher training at post-teacher training and delivery of the SEED curriculum for children at post-intervention. Another focus group interviews will be conducted with SEED trainers to get information about teachers' participation rate in the training session.
  Interventions: Behavioral: Social, Emotional, and Ethical Development (SEED) curriculum
- Waitlist control group (No Intervention): One kindergarten will be assigned to the waitlist control condition. Teachers in the waitlist control schools will wait for at least 12 weeks before they receive the training, and children in the waitlist control group will receive SEED curriculum after the teachers' training. Upon informed consent from the school principals and parents, parents, teachers, and children will also complete pre- and post-test assessments.

INTERVENTIONS:
Behavioral: Social, Emotional, and Ethical Development (SEED) curriculum — In response to fulfilling children's urgent psychosocial needs, the Bodhi Love Foundation (BLF) adapted the Kindness Curriculum for young children in Hong Kong by translating it from English to Chinese and adapting its length and content for implementation in the local kindergarten context. The adapted Kindness Curriculum, renamed as Social, Emotional, and Ethical Development curriculum (SEED), is a two-part program involving teacher training and delivery of SEED. The teacher training is consist of a 12-hour mindfulness course and a 1-day (6 hours) workshop to get familiarized with the understanding and practice of mindfulness, and the details of the SEED Curriculum. The SEED Curriculum involves 8 short sessions of basic techniques in mindfulness with 10 minutes each. In addition, it has 12 mindfulness-based lessons with specific themes for children in K2 and K3. Each lesson lasts for approximately 30-40 minutes.
  Arms: Social, Emotional, and Ethical Development (SEED) curriculum

SUMMARY:
The objectives of the present study are to (1) evaluate the feasibility and effectiveness in implementing teachers' training on mindfulness and developing their competency in delivering the Social, Emotional, and Ethical Development (SEED) curriculum to preschool children and (2) pilot the SEED curriculum at kindergartens to assess its effectiveness.

To investigate the feasibility of SEED teacher training and the SEED Curriculum, randomized controlled trials will be conducted. A minimum of two kindergartens will be recruited to participate in the study. Half of the kindergartens, teachers, and children will receive the training and SEED curriculum, while the other half will be assigned to the waitlist control condition. Upon informed consent from the school principals and parents, parents, teachers, and children will complete pre- and post-assessments, additional follow-up assessments will be conducted in intervention group. Focus group interviews will be conducted with teachers to understand their acceptability, demand, practicality, integration, and efficacy of the teacher training at post-teacher training and delivery of the SEED curriculum for children at post-intervention. Another focus group interviews will be conducted with SEED trainers to get information about teachers' participation rate in the training session.

DETAILED DESCRIPTION:
According to the World Health Organization, early child development lays a critical foundation for healthy habits and long-term development, including health and well-being, as well as changing the trajectory of the next generation in maximizing human potential. Specifically, social emotional learning (SEL) in early childhood lays the foundation for their later adjustment, including better emotional wellness and fewer internalizing and externalizing problems. Recently, numerous SEL programs have been developed worldwide . Among these evidence-based SEL programs, the Kindness Curriculum is a secular mindfulness-based SEL program designed for children between 4-6 years of age.

In Hong Kong, the Kindergarten Education Curriculum Guide has identified affective and social development as a major objective in early childhood. Better social emotional competence is associated with preschool-aged children's lower anxiety and fewer aggressive behaviors in Hong Kong. However, the implementation of evidence-based SEL programs remains immature, with very few programs available for kindergartens and kindergarten-cum-child care settings and none being mindfulness-based. In response to fulfilling children's psychosocial needs, the Bodhi Love Foundation (BLF) has adapted the Kindness Curriculum for young children in Hong Kong. With concerted efforts of a team of qualified local mindfulness teachers and Prof. Daniel Goleman as the advisor, the curriculum was translated from English to Chinese and has been adapted for implementation in the local cultural context. The adapted Kindness Curriculum, renamed as Social, Emotional, Ethical Development Curriculum (SEED), is a two-part program involving training teachers on mindfulness and delivery of SEED to young children. As such, the curriculum may be beneficial for both teachers and children.

The project's significance is to cultivate mindfulness and loving kindness among our teachers and children so to equip them with the mindset and skills needed for self-care and promotion of mental well-being. Such well-being promotion and distress prevention approach that starts early in childhood lays a critical cornerstone for children to develop healthily, which can potentially reduce the incidence of mental illness among younger generations.

ELIGIBILITY:
Inclusion Criteria:

* For children: aged 3-7 years old, understand Cantonese
* For parents: aged 18 years old or above, understand Cantonese
* For teachers: aged 18 years old or above, understand Cantonese, currently working at a kindergarten

Exclusion Criteria:

* Cannot understand Cantonese

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2023-09-16 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Mindfulness in Teaching Scale(MTS) | 8th week
  The 14-item Mindfulness in Teaching Scale(MTS) will be used to assess the extent to which teachers are consciously aware of various classroom and student activities. It contains 2 subscales measuring teacher intrapersonal and interpersonal mindfulness. Items are answered on a 5-point Likert scale (from 1 = never, to 5 = always). The total score of each dimension is obtained by summing the respective items, with higher scores indicating greater levels of Teacher Intrapersonal Mindfulness (ranging from 9 to 45) and Teacher Interpersonal Mindfulness (ranging from 5 to 25).
Mindfulness in Teaching Scale(MTS) | 12th week
  The 14-item Mindfulness in Teaching Scale(MTS) will be used to assess the extent to which teachers are consciously aware of various classroom and student activities. It contains 2 subscales measuring teacher intrapersonal and interpersonal mindfulness. Items are answered on a 5-point Likert scale (from 1 = never, to 5 = always). The total score of each dimension is obtained by summing the respective items, with higher scores indicating greater levels of Teacher Intrapersonal Mindfulness (ranging from 9 to 45) and Teacher Interpersonal Mindfulness (ranging from 5 to 25).
Copenhagen Burnout Inventory | 8th week
  The personal burnout and work-related burnout subscale in Copenhagen Burnout Inventory (CBI) will be used to measure teachers' burnout in three domains: and client-related burnout. CBI shows good reliability for each subscale (Cronbach's alpha = .85-.87).
Copenhagen Burnout Inventory | 12th week
  The personal burnout and work-related burnout subscale in Copenhagen Burnout Inventory (CBI) will be used to measure teachers' burnout in three domains: and client-related burnout. CBI shows good reliability for each subscale (Cronbach's alpha = .85-.87).
The Impermanence Awareness and Acceptance Scale | 8th week
  The 13-item Impermanence Awareness and Acceptance Scale (IMAAS) measures changes in an individual's state levels of impermanence awareness and impermanence acceptance on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).
The Impermanence Awareness and Acceptance Scale | 12th week
  The 13-item Impermanence Awareness and Acceptance Scale (IMAAS) measures changes in an individual's state levels of impermanence awareness and impermanence acceptance on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).
Interconnectedness Scale | 8th week
  The 12-item Interconnectedness Scale will be used to measure participants' awareness on their interdependent relationship with all matters in the world on a 6-point scale from 1 (totally disagree) to 6 (totally agree). The scale measures interconnectedness in three dimensions: emotional response to interconnectedness, appreciation of interconnectedness on self-development, and interconnectedness in social relations.
Interconnectedness Scale | 12th week
  The 12-item Interconnectedness Scale will be used to measure participants' awareness on their interdependent relationship with all matters in the world on a 6-point scale from 1 (totally disagree) to 6 (totally agree). The scale measures interconnectedness in three dimensions: emotional response to interconnectedness, appreciation of interconnectedness on self-development, and interconnectedness in social relations.
Mindfulness-Discernment Scale (MDS) | 8th week
  The 20-item Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) and 10-item Mindfulness subscale in the Mindfulness-Discernment Scale will be used to measure levels of mindfulness. FFMQ-SF measures five dimensions of mindfulness including observing, describing, acting with awareness, nonjudging, and nonreactivity (Baer et al., 2008) on a 5-point Likert scale ranging from 1 (never) to 5 (always). Discernment will be assessed using the 14-item Discernment subscale in the Mindfulness-Discernment Scale. Items are rated on a scale ranging from 1 (Never) to 6 (Always).
Mindfulness-Discernment Scale (MDS) | 12th week
  The 20-item Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) and 10-item Mindfulness subscale in the Mindfulness-Discernment Scale will be used to measure levels of mindfulness. FFMQ-SF measures five dimensions of mindfulness including observing, describing, acting with awareness, nonjudging, and nonreactivity (Baer et al., 2008) on a 5-point Likert scale ranging from 1 (never) to 5 (always). Discernment will be assessed using the 14-item Discernment subscale in the Mindfulness-Discernment Scale. Items are rated on a scale ranging from 1 (Never) to 6 (Always).
Nonattachment Scale(NAS)-Short Form | 8th week
  The 8-item Nonattachment Scale Short Form will be used to assess participants' flexibility and balanced approach towards life experiences on a 6-point scale. Participants rated the items from 1 (disagree strongly) to 6 (agree strongly). Three items were reversed-coded and higher scores indicate higher level of nonattachment. This abridged version was developed and validated using item response theory in Hong Kong Chinese sample.
Nonattachment Scale(NAS)-Short Form | 12th week
  The 8-item Nonattachment Scale Short Form will be used to assess participants' flexibility and balanced approach towards life experiences on a 6-point scale. Participants rated the items from 1 (disagree strongly) to 6 (agree strongly). Three items were reversed-coded and higher scores indicate higher level of nonattachment. This abridged version was developed and validated using item response theory in Hong Kong Chinese sample.
Santa Clara Brief Compassion Scale | 8th week
  The Santa Clara Brief Compassion Scale (SCBCS) is a 5-item inventory that measures compassion for others using a 7-point Likert-like scale (1 = not at all true of me to 7= very true of me), which yields a possible range of 5 to 35 points, with higher scores mean a higher level of compassion.
Santa Clara Brief Compassion Scale | 12th week
  The Santa Clara Brief Compassion Scale (SCBCS) is a 5-item inventory that measures compassion for others using a 7-point Likert-like scale (1 = not at all true of me to 7= very true of me), which yields a possible range of 5 to 35 points, with higher scores mean a higher level of compassion.
The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | 8th week
  Warwick-Edinburgh Mental Wellbeing Scale-Short is a 7-item self-report measure of subjective mental well-being on a 5-point Likert scale (1=none of the time, 5=all of the time), giving a minimum score of 14 and maximum score of 70. A higher WEMWBS score therefore indicates a higher level of mental well-being. The Chinese translation has demonstrated high levels of internal consistency, test-retest reliability, and construct validity in both community and clinical samples.
The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | 12th week
  Warwick-Edinburgh Mental Wellbeing Scale-Short is a 7-item self-report measure of subjective mental well-being on a 5-point Likert scale (1=none of the time, 5=all of the time), giving a minimum score of 14 and maximum score of 70. A higher WEMWBS score therefore indicates a higher level of mental well-being. The Chinese translation has demonstrated high levels of internal consistency, test-retest reliability, and construct validity in both community and clinical samples.
Delay of Shared Gratification Task | 8th week
  The 5-minute Delay of Shared Gratification Task measures children's sharing behavior involving the small stickers. Children will be asked to share 1-2 stickers with other people over four instances, such as sharing with cost, sharing without cost, and delay of sharing.
Delay of Shared Gratification Task | 12th week
  The 5-minute Delay of Shared Gratification Task measures children's sharing behavior involving the small stickers. Children will be asked to share 1-2 stickers with other people over four instances, such as sharing with cost, sharing without cost, and delay of sharing.
Head-Toe-Knees-Shoulders task (HTKS) | 8th week
  The 10-minute Head-Toe-Knees-Shoulders task (HTKS) measures children's behavioral regulation. Specifically, the task requires children to do the opposite of commands. For each command, the experimenter uses a 3-point scale to record the child's responses at 0 = incorrect, 1 = self-correct, and 2 = correct.
Head-Toe-Knees-Shoulders task (HTKS) | 12th week
  The 10-minute Head-Toe-Knees-Shoulders task (HTKS) measures children's behavioral regulation. Specifically, the task requires children to do the opposite of commands. For each command, the experimenter uses a 3-point scale to record the child's responses at 0 = incorrect, 1 = self-correct, and 2 = correct.
Disappointing Gift Task | 8th week
  Disappointing Gift Task measures children's emotion regulation. Specifically, they are informed that they will receive a very nice gift but end up receiving an undesirable gift, e.g., trash paper. Children's facial expression will be observed and coded based on Saarni's (1984) emotion coding system.
Strengths and Difficulties Questionnaire (SDQ) | 8th week
  A 20-item internalizing and externalizing problems subscales of the Strengths and Difficulties Questionnaire will be used to access their child's adjustment difficulties on a 3-point scale ranging from 1 (not true) to 3 (certainly true). The internalizing problems subscale capture emotional symptoms and peer relationship problems, whereas the externalizing problems subscale capture conduct problems and hyperactivity/inattention.
Strengths and Difficulties Questionnaire (SDQ) | 12th week
  A 20-item internalizing and externalizing problems subscales of the Strengths and Difficulties Questionnaire will be used to access their child's adjustment difficulties on a 3-point scale ranging from 1 (not true) to 3 (certainly true). The internalizing problems subscale capture emotional symptoms and peer relationship problems, whereas the externalizing problems subscale capture conduct problems and hyperactivity/inattention.
Social Skills Improvement System-Rating Scales (Preschool Parents version) (SSIS - SEL) | 8th week
  The SSIS SEL consists of 20 items which assess children's skills in each of the five social-emotional learning competencies: Self-Awareness, Self-Management, Social Awareness, Relationship Skills, Responsible Decision Making.
Social Skills Improvement System-Rating Scales (Preschool Parents version) (SSIS - SEL) | 12th week
  The SSIS SEL consists of 20 items which assess children's skills in each of the five social-emotional learning competencies: Self-Awareness, Self-Management, Social Awareness, Relationship Skills, Responsible Decision Making.
Behaviour Rating Inventory of Executive Function-Preschool Version | 8th week
  A 63-item Behaviour Rating Inventory of Executive Function-Preschool Version will be used to assess their child's behavioral regulation on a 3-point scale ranging from 1 (never) to 3 (often)., including inhibition, shifting, emotional control, working memory, and planning/organizing.
Behaviour Rating Inventory of Executive Function-Preschool Version | 12th week
  A 63-item Behaviour Rating Inventory of Executive Function-Preschool Version will be used to assess their child's behavioral regulation on a 3-point scale ranging from 1 (never) to 3 (often)., including inhibition, shifting, emotional control, working memory, and planning/organizing.
Children's Behavioral Questionnaire(CBQ) age 3-7-Short Form | 8th week
  In the CBQ, parents are asked to rate their child on a 7-point scale ranging from 1 (extremely untrue of your child) to 7 (extremely true of your child). Parents are also provided with a Not Applicable response option when the child has not been observed in the situation described. The standard form consists 15 subscales, in this study, 3 subscales (18 items in total) from short form are used, namely Attentional Control, Impulsivity, and Inhibitory Control. A higher score on each subscale reflects a greater level of attentional control, Impulsivity, and Inhibitory Control, respectively.
Children's Behavioral Questionnaire(CBQ) age 3-7-Short Form | 12th week
  In the CBQ, parents are asked to rate their child on a 7-point scale ranging from 1 (extremely untrue of your child) to 7 (extremely true of your child). Parents are also provided with a Not Applicable response option when the child has not been observed in the situation described. The standard form consists 15 subscales, in this study, 3 subscales (18 items in total) from short form are used, namely Attentional Control, Impulsivity, and Inhibitory Control. A higher score on each subscale reflects a greater level of attentional control, Impulsivity, and Inhibitory Control, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Winnie WS Mak, Principal Investigator — Chinese University of Hong Kong; Rebecca YM Cheung, Principal Investigator — Xi'an Jiaotong-Liverpool University
Locations (1):
- Dept of Psychology, CUHK, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blewitt C, Fuller-Tyszkiewicz M, Nolan A, Bergmeier H, Vicary D, Huang T, McCabe P, McKay T, Skouteris H. Social and Emotional Learning Associated With Universal Curriculum-Based Interventions in Early Childhood Education and Care Centers: A Systematic Review and Meta-analysis. JAMA Netw Open. 2018 Dec 7;1(8):e185727. doi: 10.1001/jamanetworkopen.2018.5727. PMID 30646283
- [Background] Bornstein MH, Hahn CS, Haynes OM. Social competence, externalizing, and internalizing behavioral adjustment from early childhood through early adolescence: developmental cascades. Dev Psychopathol. 2010 Nov;22(4):717-35. doi: 10.1017/S0954579410000416. PMID 20883577
- [Background] Collaborative for Academic, Social, and Emotional Learning (CASEL). (2021). CASEL's SEL Framework. https://casel.org/casel-sel-framework-11-2020/
- [Background] Curriculum Development Council, Education Bureau, Hong Kong SAR. (2017). Kindergarten education curriculum guide: Joyful learning through play balanced development all the way. https://www.edb.gov.hk/attachment/en/curriculum-development/major-level-of-edu/preprimary/ENG_KGECG_2017.pdf
- [Background] Dunning D, Tudor K, Radley L, Dalrymple N, Funk J, Vainre M, Ford T, Montero-Marin J, Kuyken W, Dalgleish T. Do mindfulness-based programmes improve the cognitive skills, behaviour and mental health of children and adolescents? An updated meta-analysis of randomised controlled trials. Evid Based Ment Health. 2022 Jul 12;25(3):135-42. doi: 10.1136/ebmental-2022-300464. Online ahead of print. PMID 35820989
- [Background] Flook L, Goldberg SB, Pinger L, Bonus K, Davidson RJ. Mindfulness for teachers: A pilot study to assess effects on stress, burnout and teaching efficacy. Mind Brain Educ. 2013 Sep;7(3):10.1111/mbe.12026. doi: 10.1111/mbe.12026. PMID 24324528
- [Background] Flook L, Goldberg SB, Pinger L, Davidson RJ. Promoting prosocial behavior and self-regulatory skills in preschool children through a mindfulness-based Kindness Curriculum. Dev Psychol. 2015 Jan;51(1):44-51. doi: 10.1037/a0038256. Epub 2014 Nov 10. PMID 25383689
- [Background] Heckman, J. J. (2011). The economics of inequality: The value of early childhood education. American Educator, 35(1), 31.
- [Background] Hong Kong Professional Teachers' Union. (2018, September 2). Teachers' Stress Survey. Retrieved February 15, 2023. https://hkps-dcp.org.hk/images/ourworks/TeacherStressSurveyPressRelease20180902.pdf
- [Background] Kim, S., Crooks, C. V., Bax, K., & Shokoohi, M. (2021). Impact of trauma-informed training and mindfulness-based social-emotional learning program on teacher attitudes and burnout: A mixed-methods study. School mental health, 13(1), 55-68. https://doi.org/10.1007/s12310-020-09406-6
- [Background] Lam, L. T., & Wong, E. M. (2017). Enhancing social-emotional well-being in young children through improving teachers' social-emotional competence and curriculum design in Hong Kong. International Journal of Child Care and Education Policy, 11(1), 1-14. https://doi.org/10.1186/s40723-017-0031-0
- [Background] Roeser, R. W., Skinner, E., Beers, J., & Jennings, P. A. (2012). Mindfulness training and teachers' professional development: An emerging area of research and practice. Child development perspectives, 6(2), 167-173. https://doi.org/10.1111/j.1750-8606.2012.00238.x
- [Background] Unicef. (2021, October 15). State of the world's children, caring for children's mental health. Retrieved February 15, 2023. https://webuat.unicef.org.hk/en/news/latest_news/state-of-the-worlds-children-caring-for-childrens-mental-health/
- [Background] World Health Organization. (2018). United Nations Children's Fund, World Bank Group. Nurturing care for early childhood development: a framework for helping children survive and thrive to transform health and human potential. Geneva: World Health Organization. https://apps.who.int/iris/bitstream/handle/10665/272603/9789241514064-eng.pdf